CLINICAL TRIAL: NCT02274935
Title: Cognitive Motor Interference Rehabilitation in Persons With Multiple Sclerosis
Acronym: DUETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Jacob Sosnoff, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15002
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait and balance exercise (Experimental): Traditional exercises focusing on gait and balance
  Interventions: Other: Exercise
- Cognitive training and physical exercise (Experimental): Gait and balance exercises done in combination with cognitive training (i.e. counting backwards by 7s from 98)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Balance and gait exercise twice a week for an hour
  Other Names: Physical Rehabilitation

SUMMARY:
This study examines the effect of balance and walking exercise on cognition and mobility in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
Walking and cognitive impairments are common in persons with multiple sclerosis (MS). Approximately 85% of persons with MS report walking as a major limitation, whereas 65% experience cognitive dysfunction. Traditionally, walking and cognition have been viewed as unrelated, but there is evidence of cognitive-motor interference (CMI). CMI is believed to stem from damage to common neural tracts. Recent evidence supports cognitive-motor interference in persons with MS. For example, there is evidence that walking performance declines when performed in conjunction with a simultaneous cognitive task (i.e., dual task cost [DTC] of walking) and this decline in walking performance is greater in persons with MS compared to healthy controls. This elevated cognitive-motor interference during walking is mainly associated with walking performance in persons with MS although cognitive function does play a role. Cognitive-motor interference during mobility tasks is of practical and clinical importance because it has been linked to decreased community mobility and a greater risk of falls in other clinical populations. Despite the adverse consequences of elevated CMI there is ambiguity concerning prevention and rehabilitation strategies for cognitive-motor interference in individuals with MS.

This study seeks to examine whether single and/or targeted dual task rehabilitation has a beneficial effect on CMI in individuals with MS. The results of this investigation will provide the foundation for future rehabilitation-based randomized control trials seeking to improve walking and cognitive function in persons with MS.

ELIGIBILITY:
Inclusion Criteria:Physician diagnosed MS, relapse free for 30 days, self reporting problems with multitasking -

Exclusion Criteria:We will exclude all individuals with risk factors contra-indicative for undertaking strenuous exercise. Participants will verbally respond to a health history questionnaire. Those individuals who are asymptomatic and meet no more than one risk factor threshold including family history of coronary heart disease, cigarette smoking, hypertension, high cholesterol, diabetes, obesity, and sedentary lifestyle will be considered at low risk and included for participation.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cognitive Motor interference | 12 weeks
  This will be operationalized as the percent change in walking velocity from single (walking only) to dual task (walking while thinking). Participants will complete a total of 8 walking trials over a 20' pressure sensitive (Zeno™) walkway. Four at a comfortable walking speed and four as fast as possible. Half of the trials at each speed will be conducted while reciting every other letter of the alphabet (i.e. N, P, R, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosnoff, PhD, Principal Investigator — Associate Professor, University of Illinois
Locations (1):
- Motor control research lab, Urbana, Illinois, United States